CLINICAL TRIAL: NCT01948570
Title: Clinical Study for the Evaluation of P-3075 Cream on Acne Treatment
Acronym: ANTI-ACNE
Status: Completed | Type: Observational
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Dermatologist, Derming SRL
Other Study IDs: E0113
Record Dates: First submitted 2013-09-06; First posted 2013-09-23 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2013-09

CONDITIONS: Acne
Keywords: acne,comedones, oily skin
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- not in therapy (GROUP 1): A fixed quantity of the medical device will be applied on the face twice a day, in the morning and in the evening (always at the same hour), with a mild massage according to the instructions received by the investigator during the baseline visit (T0).
- in therapy (GROUP 2): A fixed quantity of the medical device will be applied on the face twice a day, in the morning and in the evening (always at the same hour), with a mild massage according to the instructions received by the investigator during the baseline visit (T0). Group 2 will continue also the standardised treatment with topical or systemic retinoids, benzoyl peroxide, clindamycin or AHA until the end of the study

SUMMARY:
Primary end point of the study is the clinical and non-invasive instrumental evaluation of the activity of P-3075 cream on subjects with acne: 20 subjects with a mild/moderate grade and 20 subjects with a moderately severe/severe grade, according to Cunliffe' classification.

Secondary end-points are the cosmetic acceptability and efficacy evaluation by the volunteers and the local tolerability assessed by the investigator and the subjects.

DETAILED DESCRIPTION:
This is an open controlled clinical trial. The product will be applied for a period of 4 weeks and 3 visits will be performed: a baseline visit (T0), an intermediate visit after 2 weeks (T2) and a final visit after 4 week-treatment (T4).

The subjects will be enrolled and divided in 2 groups according to their acne grade (20 subjects with mild/moderate grade and 20 subjects with moderately severe/severe), a concomitant therapy is allowed only for volunteers with acne moderately severe/severe.

Each volunteer, fulfilling the inclusion criteria, will perform a cosmetic treatment with the study product on all the face, for 4 weeks.

A fixed quantity of the medical device will be applied on the face twice a day, in the morning and in the evening (always at the same hour), with a mild massage according to the instructions received by the investigator during the baseline visit (T0). Group 2 will continue also the standardised treatment with topical or systemic retinoids, benzoyl peroxide, clindamycin or AHA until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* both genders;
* age > 16 years old;
* acne of mild/moderate grade, not in therapy (GROUP 1);
* acne of moderately severe/severe grade, in therapy with topical or systemic retinoids, benzoyl peroxide, clindamycin or AHA (GROUP 2);
* accepting to follow the instructions received by the investigator;
* available to return to the study centre at the protocol visits;
* accepting to not change the normal life habits regarding: food, physical activity, face cleansing;
* accepting not to receive any other drug/cosmetic treatment able to interfere with the study results;
* accepting to sign the informed consent form (under 18 years the signature of both parents is required).

Exclusion Criteria:

* Pregnancy (only for female subjects) - for subjects belonging to Group 2, a control pregnancy test could be required at T2 and T4 in case of assumption of an anti-acne drug with potential teratogenic effects; these subjects must confirm to use adequate contraceptive precautions in order to avoid pregnancies;
* lactation (only for female subjects);
* subjects whose insufficient adhesion to the study protocol is expected;
* subjects who changed the anti-acne therapy during the 2 months prior to the study inclusion;
* concomitant participation in other studies or in the last 3 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on volunteers of both genders, aged > 16 years old: 20 subjects presenting acne of mild/moderate grade not in therapy (GROUP 1) and 20 subjects presenting acne of moderately severe/severe grade in therapy with topical or systemic retinoids, benzoyl peroxide, clindamycin or AHA (GROUP 2).
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
clinical and non-invasive instrumental evaluation of the activity of P-3075 cream on subjects with acne | 1 month
  Visual evaluations (comedones, dryness, desquamation, papules, pustoles, microcystis) Tissue dielectric constant (superficial and deep hydration), sebumetry and optical colorimetry (skin colour), follicular biopsy, sebutape image analysis

SECONDARY OUTCOMES:
subjects' self assessment | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Adele Sparavigna, Physician, Principal Investigator — Derming SRL
Locations (1):
- DermIng S.r.l, Monza, MB, Italy

REFERENCES:
- [Background] Adityan B, Kumari R, Thappa DM. Scoring systems in acne vulgaris. Indian J Dermatol Venereol Leprol. 2009 May-Jun;75(3):323-6. doi: 10.4103/0378-6323.51258. No abstract available. PMID 19439902
- [Background] Alanen E, Lahtinen T, Nuutinen J. Penetration of electromagnetic fields of an open-ended coaxial probe between 1 MHz and 1 GHz in dielectric skin measurements. Phys Med Biol. 1999 Jul;44(7):N169-76. doi: 10.1088/0031-9155/44/7/404. PMID 10442720
- [Background] Becker W.D., Bajor J.S., Hoyberg K., Hillmer S., Thibouto D., Knaggs H. Measurement Of Human Surface Sebum Levels The Journal of Investigative Dermatology, Vol. 110, No. 4, April 1998
- [Background] Clarys P.M., Barel A.O. Sebumetry: A comparison between Lipid Collection Techniques. Skin Research and Technology, Vol.2, No.4, Nov.1996
- [Background] Cunliffe WJ, Shuster S. The rate of sebum excretion in man. Br J Dermatol. 1969 Sep;81(9):697-704. doi: 10.1111/j.1365-2133.1969.tb16211.x. No abstract available. PMID 4243403
- [Background] Curry AS, Gettings SD, McEwen GN CTFA safety testing guidelines. The Cosmetic, Toiletry and Fragrance Association, Washington, (1991)
- [Background] Elsner P. Sebum Bioengineering of the Skin: Methods and Instrumentation, CRC Press 1995
- [Background] Fernay, Voltaire The World Medical Association (1989) "World Medical Association Declaration of Helsinki", Hong-Kong
- [Background] ICH Harmonised Tripartite Guideline - Guideline for Good Clinical Practice International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use: May 1996
- [Background] Kiiskinen M., Nuutinen J. and Alanen E. Measurement depths of a skin-water analyzer (MoistureMeter D) Skin Res Technol, Vol 11: 292, 2005
- [Background] Klingman A.M., Miller D.L., McGinley K.J. Sebutape: A device for visualizing and measuring human sebaceous secretion. J. Soc. Cosmet. Chem. 37:369-374, 1896
- [Background] Lahtinen, T., Nuutinen, J., Alanen, E. Dielectric properties of the skin In: Radio Frequency Radiation Dosimetry. Editors: B. J. Klauenberg and D. Miklavcic. Kluwer Academic Publishers, the Netherlands, 2000
- [Background] Lahtinen T, Nuutinen J, Alanen E. Dielectric properties of the skin. Phys Med Biol. 1997 Jul;42(7):1471-2. doi: 10.1088/0031-9155/42/7/020. No abstract available. PMID 9253055
- [Background] Mayrovitz HN, Luis M. Spatial variations in forearm skin tissue dielectric constant. Skin Res Technol. 2010 Nov;16(4):438-43. doi: 10.1111/j.1600-0846.2010.00456.x. PMID 20923455
- [Background] Pierard GE, Pierard-Franchimont C, Le T, Lapiere C. Patterns of follicular sebum excretion rate during lifetime. Arch Dermatol Res. 1987;279 Suppl:S104-7. doi: 10.1007/BF00585931. PMID 2959210
- [Background] Rieger M.M., Battista G.W. Some experiences in the safety testing of cosmetics J. Soc. Cosmet. Chem. 15:161 -172 (1964)
- [Background] Sachs L. Applied statistics: a handbook of techniques. Heidelberg: Springer, 1981:536-539
- [Background] Sparavigna A. Un metodo di valutazione della secrezione sebacea a livello dei singoli follicoli: il Sebutape. Cosmesi Dermatologica 30: 73-75, 1990
- [Background] Thune P, Gustavsen T. Comparison of two photoelectric techniques for quantitative measurements of skin surface lipids. Acta Derm Venereol Suppl (Stockh). 1987;134:30-2. No abstract available. PMID 3481919
- [Background] Van de Vijver LPL, Boelsma E, Bausch-Goldbohm RA, Roza L. Subjective skin condition and its association with objective skin measurements. Cosm Toil 2003: 118: 45-54
- [Background] Wilhelm KP, Elsner P, Berardesca E, Maibach HI Bioengineering of the skin: Skin surface imaging and analysis. CRC Press, Boca Raton, 1997
- [Background] 9th international symposium
- See also: Investigation center — http://www.derming.com
- See also: Text sponsor — http://www.polichem.com